CLINICAL TRIAL: NCT05556304
Title: In Vivo Evaluation of Perineal Mechanical Properties During Childbirth
Acronym: MecaPer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2022/694
Record Dates: First submitted 2022-09-19; First posted 2022-09-27 (Actual); Last update posted 2022-09-27 (Actual); Status verified 2022-05

CONDITIONS: Perineum; Rupture; Perineum; Tear; Perineal Tear
Keywords: perineal tear; hyperelasticity
MeSH Terms: conditions — Rupture; Lacerations | interventions — Restraint, Physical

STUDY DESIGN:
Intervention Model Description: prospective, longitudinal and single-center study
Masking Description: The study design includes a consultation during pregnancy between 36 and 38 weeks of gestation and an assessment in the delivery room during childbirth
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- assessment in the 8th month of pregnancy and during delivery (Other): The study design includes a consultation during pregnancy between 36 and 38 weeks of gestation and an assessment in the delivery room during childbirth
  Interventions: Other: assessment in the 8th month of pregnancy and during delivery

INTERVENTIONS:
Other: assessment in the 8th month of pregnancy and during delivery — * Day 0: presentation of the study
  * During pregnancy between Day 0 and 36-38SA: inclusion
  * During pregnancy: collection of pelvic MRI data if performed during pregnancy for maternal or fetal reasons
  * Between 36 and 38 WG: collection of demographic, obstetrical, fetal ultrasound and clinical data / Perineal elastographic recording / Recording of the perineal deformation by stereovision camera
  * In the delivery room, at the beginning of labor and before pushing: collection of clinical data / Collection of obstetrical ultrasound data / Perineal elastographic recordings / Recording of the perineal deformation by stereovision camera
  * In the delivery room, during expulsion : recording of the perineal deformation by stereovision camera
  * In the delivery room, after childbirth: collection of obstetrical, clinical and neonatal data / Perineal elastographic recordings / Cephalic and shoulder measurements of the newborn with a tape measure

SUMMARY:
The objective of this work is to evaluate perineal elasticity and deformation and the perineal stresses induced by the fetus during delivery.

DETAILED DESCRIPTION:
The objective of this work is to evaluate perineal elasticity and deformation and the perineal stresses induced by the fetus during delivery.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant and volunteer women >18 years old
* Primiparous
* With a singleton pregnancy
* No objection from the subject and the spouse to participate in the study

Exclusion Criteria:

* History of prior delivery or c-section
* History of perineal troubles
* BMI > à 35 mg/m²
* History of chronic muscular disease or connective tissue pathology
* Psychiatric pathology requiring hospitalization
* Patients who do not understand the French language
* Legal incapacity or limited legal capacity
* Patients unlikely to cooperate

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-10-01 (Estimated); Primary Completion 2022-12-01 (Estimated); Study Completion 2023-10-30 (Estimated)

PRIMARY OUTCOMES:
maximum value of equivalent deformation obtained by stereovision camera | delivery
  maximum value of equivalent deformation obtained by stereovision camera

SECONDARY OUTCOMES:
Delta between the minimum and maximum width of GH, and between the maximum and minimum length of PB | pregnancy
  Delta between the minimum and maximum width of GH, and between the maximum and minimum length of PB
Delta between the minimum and maximum width of GH, and between the maximum and minimum length of PB | delivery
  elta between the minimum and maximum width of GH, and between the maximum and minimum length of PB
Correlation between perineal deformation values and perineal tears | delivery
  Correlation between perineal deformation values and perineal tears
Correlation between perineal deformation values and fetal parameters | pregnancy
  Correlation between perineal deformation values and fetal parameters
Correlation between perineal deformation values and fetal parameters | delivery
  Correlation between perineal deformation values and fetal parameters
Correlation between fetal ultrasound and neonatal parameters and perineal tears | delivery
  Correlation between fetal ultrasound and neonatal parameters and perineal tears
Evolution of the elasticity of the perineal body and the SAE during delivery | delivery
  Evolution of the elasticity of the perineal body and the SAE during delivery
Correlation between elasticity of the perineal body and perineal tears | pregnancy
  Correlation between elasticity of the perineal body and perineal tears
Correlation between elasticity of the perineal body and perineal tears | delivery
  Correlation between elasticity of the perineal body and perineal tears
Correlation between the elasticity of the external anal sphincter and perineal tears | pregnancy
  Correlation between the elasticity of the external anal sphincter and perineal tears
Correlation between the elasticity of the external anal sphincter and perineal tears | delivery
  Correlation between the elasticity of the external anal sphincter and perineal tears

REFERENCES:
- [Derived] Lallemant M, Kadiake T, Lejeune A, Cosson M, Chambert J, Jacquet E, Mottet N. Perineal body and anal sphincter biometrics and stiffness using elastography during labor: a feasibility study. Eur J Obstet Gynecol Reprod Biol. 2025 May;309:48-54. doi: 10.1016/j.ejogrb.2025.03.034. Epub 2025 Mar 12. PMID 40107173
- [Derived] Lallemant M, Kadiake T, Lejeune A, Cosson M, Chambert J, Jacquet E, Mottet N. Exploring the influence of perineal biometrics and stiffness measured by elastography during pregnancy on perineal tears : A pilot study. J Gynecol Obstet Hum Reprod. 2025 Mar;54(3):102904. doi: 10.1016/j.jogoh.2025.102904. Epub 2025 Jan 11. PMID 39805482